CLINICAL TRIAL: NCT06783361
Title: Accelerated Transcranial Magnetic Stimulation in Treatment-Resistant Depressed Patients: Comparison Of The Effectiveness Of Bilateral Theta Bursts With Unilateral Theta Bursts
Brief Title: Accelerated Transcranial Magnetic Stimulation in Treatment-Resistant Depressed Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Omer Faruk Uygur, associate professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-04/10; Atatürk University (Other: Scientific Research Projects Coordination Unit)
Record Dates: First submitted 2024-12-13; First posted 2025-01-20 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Treatment Resistant Depression (TRD); Transcranial Magnetic Stimulation; Accelerated Protocol; Sham-controlled; Bilateral rTMS; Unipolar Major Depressive Disorder
Keywords: treatment resistant depression; non-invasive brain stimulation; transcranial magnetic stimulation; sham controled; unipolar major depressive disorder
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A group (Active Comparator): iTBS with eight digit coils to the left dorsolateral prefrontal cortex and cTBS with a figure-of-eight coil to the right dorsolateral prefrontal cortex.
  Interventions: Device: Transcranial Magnetic Stimulation with figure-eight coil
- B group (Sham Comparator): iTBS with eight digit coils to the left dorsolateral prefrontal cortex and sham Sham cTBS with a figure-of-eight coil to the right dorsolateral prefrontal cortex.
  The sham cTBS treatment will be administered by placing the coil at a 45-degree angle to the application site.
  Interventions: Device: Transcranial Magnetic Stimulation with figure-eight coil

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation with figure-eight coil — A total of 50 sessions will be applied for 2 weeks, 5 sessions a day, 5 days a week. There will be at least 30 minutes rest time between each session. It includes first an intermittent theta burst (iTBS) protocol at a frequency of 5 Hz with 1800 pulses to the left DLPFC at 90% motor threshold, followed by a continuous theta burst (cTBS) protocol at a frequency of 5 Hz with 600 pulses to the right DLPFC at 80% motor threshold.
  Other Names: active treatment
  Arms: A group
Device: Transcranial Magnetic Stimulation with figure-eight coil — A total of 50 sessions will be applied for 2 weeks, 5 sessions a day, 5 days a week. There will be at least 30 minutes rest time between each session. One session will consist of a high frequency (5 Hz) intermittent theta burst (iTBS) of 1800 pulses at 90% motor threshold to the left DLPFC followed by a pseudo continuous theta burst (cTBS) of 600 pulses at 5 Hz frequency at 80% motor threshold to the right DLPFC. The sham cTBS treatment will be applied by placing the coil at a 45-degree angle to the application site.
  Other Names: sham control group
  Arms: B group

SUMMARY:
Depression is the leading cause of disability worldwide and around 800,000 suicides occur each year. According to the World Health Organization, major depressive disorder (MDD) is expected to be the leading cause of the global burden of disease by 2030. One third of MDD patients do not respond to first-line pharmacologic and psychotherapeutic antidepressant treatments. New antidepressant treatments that are safe, tolerable, fast-acting, durable and effective are needed. Transcranial magnetic stimulation (TMS) is a promising form of non-invasive brain stimulation with rapid antidepressant and suicide prevention effects in MDD. TMS applied to the left dorsolateral prefrontal cortex (DLPFC) is a non-invasive brain stimulation technique approved by the US Food and Drug Administration (FDA) for treatment-resistant depression. TMS involves passing an electric current through a magnetic coil placed on the surface of the scalp, producing a high-intensity magnetic field that travels through the scalp, skull and meninges, stimulating neuronal tissue. This in turn causes changes in functional connectivity. The mechanism of TMS on core depressive symptoms is hypothesized to be mediated in part through indirect inhibitory functional connectivity from the left DLPFC to the subgenual anterior cingulate cortex (sgACC).

DETAILED DESCRIPTION:
The aim of this study was to investigate whether recurrent TMS (rTMS) and theta burst stimulation (TBS) are superior to each other when applied unilaterally and bilaterally in treatment-resistant MDD. As stated in the reference articles, a similar study was conducted unilaterally at Stanford University and achieved 70% remission rates. Our goal is that bilateral administration will result in longer treatment compliance and duration of effect compared to unilateral administration. This study aims to monitor the change in neurocognitive functions of patients with moderate to severe depression diagnosed with major depression according to DSM 5 criteria, whose treatment is prescribed by their physician as transcranial magnetic stimulation (TMS) and whose current pharmacological treatment is continued concurrently with TMS treatment, at the controls to be performed before TMS treatment, 1 week, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks and 14 weeks after the start of TMS treatment. For this purpose, structured neuropsychological tests with Turkish validity and reliability studies will be applied to the patients. In addition, the study aims to evaluate whether there will be a decrease in the severity of depression after TMS treatment and whether there is any change in depression severity and symptoms in the 1st week, 2nd week, 4th week, 6th week, 8th week, 10th week and 14th week controls through the scales measuring the severity of depression to be applied to the patients participating in the study.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years old
2. Patients diagnosed with Major Depressive Disorder according to DSM 5 and the severity of their illness
3. Scoring 7 points or more on the Maudsley staging method
4. Having depression unresponsive to 2 different antidepressants
5. No clinical mental retardation
6. Agree to participate in the study
7. Hamilton Depression Rating Scale-17 [HDRS] score of 20 or higher
8. Montgomery Asberg Depression Rating Scale [MADRS] score of 20 or above
9. Being right hand dominant
10. Having used the same antidepressant at the same dose for the last 4 weeks

Exclusion Criteria:

1. Diagnosed with a neurological or metabolic disease that affects cognitive functions (Systemic diseases such as diabetes mellitus, cardiovascular disease, cerebrovascular disease, chronic renal failure, Parkinson's disease, multiple sclerosis, polyneuropathy, inflammatory rheumatologic disease and malignancies)
2. Having a foreign body such as a pacemaker, intracranial implant that can magnetically interact
3. Hearing and visual impairments that prevent communication
4. Unstable or acute medical conditions
5. Pregnancy or breastfeeding
6. Having a primary psychiatric disorder other than major depressive disorder
7. Being diagnosed with severe MDD with psychotic features

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Depression severity | pretreatment, 1 week, 2 weeks, 4 weeks, 6 weeks, 10 weeks and 14 weeks
  The Montgomery-Asberg Depression Rating Scale. The minimum and maximum scores are 0-60. Higher scores mean a worse outcome.
Depression severity | pretreatment, 1 week, 2 weeks, 4 weeks, 6 weeks, 10 weeks and 14 weeks
  The Hamilton Depression Rating Scale-17. The minimum and maximum scores are 0-51. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Anxiety severity | pretreatment, 1 week, 2 weeks, 4 weeks, 6 weeks, 10 weeks and 14 weeks
  Hamilton Anxiety Rating Scale. The minimum and maximum scores are 0-56. Higher scores mean a worse outcome.
Suicidal ideation score of The Hamilton Depression Rating Scale-17 | pretreatment, 1 week, 2 weeks, 4 weeks, 6 weeks, 10 weeks and 14 weeks
  Suicidal ideation score on the third question of the Hamilton Depression Rating Scale-17. The minimum and maximum scores are 0-4. Higher scores mean a worse outcome.
Suicidal ideation score of The Montgomery-Asberg Depression Rating Scale | pretreatment, 1 week, 2 weeks, 4 weeks, 6 weeks, 10 weeks and 14 weeks
  Suicidal ideation score on the tenth question of the Montgomery-Asberg Depression Rating Scale. Minimum and maximum scores range from 0-6. Higher scores mean a worse outcome.
Insomnia Severity | pretreatment, 2 weeks, 4 weeks, 6 weeks, 10 weeks and 14 weeks
  It is measured with the Pittsburgh Sleep Quality Index (PSQI). The minimum and maximum scores are 0-21. Higher scores mean a worse outcome.
Insomnia Severity | pretreatment, 4 weeks, 10 weeks and 14 weeks
  It is measured with the Insomnia Severity Index (ISI). The minimum and maximum scores are 0-28. Higher scores mean a worse outcome.
Cognitive Assessment | pretreatment, 4 weeks, 10 weeks and 14 weeks
  Montreal Cognitive Assessment (MoCA) : The maximum score that can be obtained from the test is 30. A total score of 21 and above indicates that the participant is within normal limits.
Functionality Severity | pretreatment, 1 week, 2 weeks, 4 weeks, 6 weeks, 10 weeks and 14 weeks
  Functioning Assessment Short Test (FAST): It is used to measure patients' functionality. The minimum and maximum scores are 0-66. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Omer Faruk UYGUR, Associate professor doctor, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No